CLINICAL TRIAL: NCT06293976
Title: Susceptibility for Entrainment: Role of Ventilator Settings on the Occurrence of Reverse Triggering and Its Physiological Consequences - the SEVeRe Study
Acronym: SEVERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4506
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-05

CONDITIONS: Respiration, Artificial; Reverse Triggering
Keywords: Hypnotics and Sedatives; Respiratory Muscles
MeSH Terms: conditions — Respiratory Aspiration | interventions — Tidal Volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients under mechanical ventilation (Experimental): Patients intubated for more than 12 hours, on assist-control ventilation, not triggering the ventilator with or without reverse triggering, exposed to sedation for at least 6 hours, with a sedation-agitation score ≤ 4.
  Interventions: Other: Changes in the ventilator respiratory rate and tidal volume

INTERVENTIONS:
Other: Changes in the ventilator respiratory rate and tidal volume — With the ventilator on volume control and Vt at 6 ml/kg of predicted body weight (PBW) (standard clinical practice), an end-expiratory occlusion of 30 seconds on the ventilator will be performed to search for intrinsic respiratory rate (RR). The set RR will be modified from 6 breaths per minute (bpm) below up to 6 bpm above the clinical RR in steps of 2 bpm every 1 minute (random order). The changes in RR described above will be repeated with Vt set at 5, 7 and 8 ml/kg PBW (random order). The steps described above will be aborted at any point if SpO2 drops below 85% for at least two minutes, mean arterial pressure drops below 60 mmHg, or plateau pressure >35 cmH2O.
  If an intrinsic respiratory rate ≥8 bpm is present and P/F ratio is ≥150, it will be propose to the clinician to place the patient in pressure support at a level preferred by clinicians for 5 minutes. If the patient tolerates well, it will be propose to the clinician to maintain the patient in pressure support ventilation,

SUMMARY:
Background: Reverse triggering (RT) is a frequent phenomenon observed in sedated patients under a mechanical ventilation mode called assist-control ventilation. RT is when the ventilator would trigger the patient's respiratory effort instead of the correct order of the patient's respiratory effort triggering the ventilator. Reverse triggering can have negative consequences (loss of protective lung ventilation, and causing double breaths - with the ventilator giving two consecutive breaths and not allowing the patient to exhale) but also offer some protective effects (avoid diaphragm disuse atrophy). The balance of its negative vs positive effects depends on its frequency and magnitude of its associated respiratory effort. Respiratory entrainment is the most often referred mechanism involving a change in patient's rate of breathing effort from that of patient's intrinsic rate to the rate of mechanical insufflation. The specific ventilatory settings associated with or responsible for RT remains unknown.

Aims: To assess in mechanically ventilated critically ill patients the influence of the set respiratory rate (RR) and tidal volume (Vt) on the presence/development of RT and to describe the pattern of respiratory muscle activity during Reverse Triggering (RT).

Methods. 30 adult patients (15 in each group), sedated and under assist-controlled ventilation will be included. Ventilator settings will be modified to modulate the frequency and magnitude of reverse triggering. Initially, with the ventilator on a mode called volume control, which means the ventilator controls the amount of air (tidal volume) and the number of breaths the patients gets every minute (respiratory rate [RR]). The tidal volume will be set at the current standard clinical practice setting (6 ml/kg of predicted body weight). The presence of an intrinsic respiratory rate will be assessed with an end-expiratory occlusion maneuver. Next, the number of breaths the ventilator gives per minute (RR) will be changed from 6 breaths less to 6 breaths more, in steps of 2 breaths every minute. The protocol will be repeated again changing the amount of air the patients gets (tidal volume) from 4, 5, 7 and 8 ml/kg. Continuous recordings of airway pressure, flow, esophageal pressure, electrical activity of the diaphragm, main accessory muscles and frontal electroencephalography will be obtained during the protocol and baseline clinical and physiological characteristics and outcomes will be recorded. A validated software will be used to detect RT and measure the intensity and timing of each muscle electrical activity and the magnitude of the inspiratory effort during RT.

DETAILED DESCRIPTION:
Participants. Critically ill patients (n: 30; aimed recruitment of equal numbers of men and women) aged 18 years or older admitted to the St. Michael's Hospital, Unity Health Toronto, Ontario, Canada.

Inclusion criteria:

* patients intubated for more than 12 hours
* exposed to sedation for at least 6 hours
* with a sedation-agitation score ≤ 4
* and corresponding to one of the following categories based on bedside inspection of ventilator waveforms:

  1. patients on assist-control ventilation having reverse triggering at clinical settings (n: 15).
  2. patients on assist-control ventilation without reverse triggering at the clinical settings (n: 15).

Exclusion criteria:

* primary severe neurological disorders
* previous lung transplant
* contraindications for esophageal catheter insertion
* current use of continuous neuromuscular blocking agents at the time of the study procedure
* severe metabolic acidosis (pH < 7.25) at the time of study procedure. Study design. Briefly, first the ventilator Vt is set at 6 ml/kg of predicted body weight (PBW) (i.e., clinical practice recommendation) and either a up to 30sec-long (or two inspiratory efforts) end-expiratory occlusion maneuver will be performed on the ventilator or the patient will be switched to pressure support for 30 - 60 sec (based on discussion with the clinical team) to assess the presence or absence of patient's intrinsic RR.

Secondly, the influence of the ventilator RR on both the occurrence of reverse triggering and the level of effort associated with the reverse triggered breath will be assessed. In random order the ventilator RR will be modified from 6 bpm below up to 6 bpm above the clinical RR in steps of 2 bpm every 1 minute (Figure 1). A 1-minute stage at the patients clinical settings of ventilation in-between each step will be performed to minimize changes in PaCO2.

Thirdly, the influence of the Vt set on the ventilator on both the occurrence of reverse triggering and the level of effort associated with the reverse triggered breath will be assessed. The ventilator Vt will be set to 5 ml/kg PBW, 7 and 8 ml/kg PBW in random order and for each volume, repeat the sequence described in the paragraph above. A 1-minute clinical settings ventilation will be performed in-between each step to minimize changes in PaCO2.

Next, the patient will be returned to their initial clinical settings. Another end-expiratory occlusion of up to 30 seconds (or two inspiratory efforts) or switch the patient to pressure support for 30 - 60 sec (based on discussion with the clinical team) will be performed to search for an intrinsic RR (i.e., intrinsic respiratory drive). If an intrinsic respiratory rate ≥8 breaths per minute is present and P/F ratio is ≥150, it will propose to the clinician to place the patient in pressure support at a level preferred by clinicians for 5 minutes. If the patient tolerates well 5 minutes in pressure support, it be will propose to the clinician to maintain the patient in pressure support ventilation.

The steps described above will be aborted at any point if SpO2 drops below 85% for at least two minutes, mean arterial pressure drops below 60 mmHg, or plateau pressure >35 cmH2O.

Additionally, the ventilator waveforms and electroencephalography (EEG) will be recorded continuously for the next 24 hours to investigate whether the presence of intrinsic RR was associated with changes in the ventilation mode by the clinician and brain activity.

ELIGIBILITY:
Inclusion criteria:

* Patients intubated for more than 12 hours
* On assist-control ventilation, not triggering the ventilator
* Exposed to sedation for at least 6 hours
* With a sedation-agitation score ≤ 4.

Exclusion Criteria:

* primary severe neurological disorders
* previous lung transplant
* contraindications for esophageal catheter insertion
* current use of continuous neuromuscular blocking agents at the time of the study procedure
* severe metabolic acidosis (pH < 7.25) at the time of study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The rate of of reverse triggered breaths occurring after each change in the ventilator respiratory rate and tidal volume. | 1 minutes
  The rate of reverse triggered breaths occurring after each change in the ventilator respiratory rate and tidal volume.
The magnitude of the effort, measured by the drop in the esophageal pressure in cmH2O, associated with the reverse triggered breaths after each change in the ventilator respiratory rate and tidal volume | 1 minute
  The magnitude of the effort, measured by the drop in the esophageal pressure in cmH2O, associated with the reverse triggered breaths after each change in the ventilator respiratory rate and tidal volume

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, Principal Investigator — Unity Health Toronto - St. Michael's Hospital
Locations (1):
- Unity Health Toronto - St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No